CLINICAL TRIAL: NCT07050615
Title: To Compare the Frequency of Post-operative Pain of Continuous Versus Interrupted Suturing Technique in Episiotomy
Brief Title: Comparison of the Frequency of Post-Operative Pain of Continuous Versus Interrupted Suturing Techniques in Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAROOJ-SITH
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous group (Experimental): In this group patients under going episiotomy, went through continuous suturing
  Interventions: Procedure: Continuous suturing
- Interrupted group (Experimental): In this group patients under going episiotomy, went through interrupted suturing
  Interventions: Procedure: Interrupted suturing

INTERVENTIONS:
Procedure: Continuous suturing — In this group, episiotomy repair was done using the continuous suturing.
  Arms: Continuous group
Procedure: Interrupted suturing — In this group, episiotomy repair was done using the interrupted suturing.
  Arms: Interrupted group

SUMMARY:
Post-operative pain is the most prevalent issue following an episiotomy, greatly affecting patients both physically and mentally, resulting in increased morbidity. This study seeks to compare the effectiveness of continuous and interrupted suturing techniques for episiotomy post-operative pain among the local population.

DETAILED DESCRIPTION:
There is a lack of recent local data regarding the management of post-operative pain using different suturing techniques. The findings of this study would help in adopting a more effective technique, resulting in reducing the postoperative pain and lowering morbidity. Practical recommendations can be made to enhance routine practices and establish guidelines for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females
* Aged 20-40years
* Undergoing an episiotomy to facilitate the delivery of the head in the labor room
* First or second pregnancy
* Gestational age of 37-41+6 weeks

Exclusion Criteria:

* Females, undergone an instrumental vaginal delivery
* With a history of previous perineal surgery
* With high-risk pregnancies (those having hypertension, anemia or bleeding tendency, diabetes mellitus, a suspected genital infection)
* With impaired immunity
* Taking corticosteroids

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 48 hours
  Post-operative pain (yes/no) was noted using the visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Arooj Akram, Principal Investigator — Shahida Islam Medical Complex, Lodhran; Joveria Sadaf, Principal Investigator — Shahida Islam Medical Complex, Lodhran
Locations (1):
- Shahida Islam Medical Complex, Lodhran, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.